CLINICAL TRIAL: NCT03810456
Title: Improving Veteran Functioning With Intensive Transdiagnostic CBT for Anxiety
Brief Title: Transdiagnostic Cognitive Behavioral Treatment for Anxiety
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2160-R; 5I01RX002160-02 (NIH)
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Results first posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2022-10

CONDITIONS: Anxiety Disorders
Keywords: Cognitive Behavior Therapy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The proposed study is a randomized controlled trial with 3 treatment arms. A transdiagnostic group CBT protocol will be compared in a compressed weekend format (iCBT) with a standard group delivery format involving 3 months of weekly sessions (sCBT). A treatment as usual (TAU) condition will be included to compare outcomes. Veterans with one or more anxiety-based disorder(s) (with or without co-occurring depression) will be randomized to one of the three treatment arms. Veterans will be asked to attend a total of four assessments during the study including a baseline evaluation, 1-month, 3-month, and 6-month follow-ups.
Who Masked: Outcomes Assessor
Masking Description: Persons completing follow-up assessments will be masked to the conditions to which patients were randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- iCBT (Active Comparator): Patients in this arm will receive transdiagnostic CBT delivered in an intensive format over one weekend.
  Interventions: Behavioral: Intensive Cognitive Behavior Therapy (iCBT)
- sCBT (Active Comparator): Patients in this arm will receive transdiagnostic CBT delivered in a standard weekly format for 12 weeks.
  Interventions: Behavioral: Standard Cognitive Behavior Therapy (sCBT)
- TAU (No Intervention): Patients in this arm will not receive transdiagnostic CBT but will receive treatment as usual.

INTERVENTIONS:
Behavioral: Intensive Cognitive Behavior Therapy (iCBT) — Participants randomized to iCBT will receive 16 hours of cognitive behavioral therapy for anxiety over one weekend. The treatment entails psychoeducation, cognitive restructuring and exposure exercises.
  Arms: iCBT
Behavioral: Standard Cognitive Behavior Therapy (sCBT) — Participants randomized to sCBT will receive 16 hours of cognitive behavioral therapy for anxiety weekly over a period of 12 weeks. The treatment entails psychoeducation, cognitive restructuring and exposure exercises.
  Arms: sCBT

SUMMARY:
This study is a randomized controlled trial examining the effectiveness of a transdiagnostic cognitive behavioral treatment (CBT) in improving Veterans' community reintegration and quality of life. Veterans with anxiety-based disorders, including posttraumatic stress, panic, social anxiety, and generalized anxiety disorders (with or without co-occurring depression) will be randomized to an intensive CBT (iCBT) treatment delivered over one weekend, standard CBT (sCBT) delivered over 12 weeks or treatment as usual (TAU). The study will also evaluate the potential of the compressed weekend format of iCBT in producing more rapid improvement in outcomes and increasing psychotherapy engagement compared with a standard psychotherapy format. Qualitative interviews will be conducted with Veterans who receive iCBT and their family members to examine how iCBT and environmental factors impacted their process of recovery.

DETAILED DESCRIPTION:
The current project proposes to evaluate a brief but intensive transdiagnostic CBT that simultaneously targets multiple anxiety disorders with or without co-occurring depression. This will be accomplished by evaluating an innovative treatment delivery method that directly addresses barriers associated with standard psychotherapy delivery. The main objectives are to (1) determine if an intensive CBT protocol (iCBT) delivered over one weekend can improve community reintegration, quality of life, and emotional functioning compared with standard CBT (sCBT) and treatment as usual (TAU); (2) examine the rates of psychotherapy engagement in iCBT compared with sCBT; and (3) obtain a deeper understanding, through qualitative interviews with Veterans and their family members, of how iCBT and environmental factors may impact the process of reintegration and quality of life.

The proposed study is a randomized controlled trial with 3 treatment arms. A transdiagnostic group CBT protocol will be compared in a compressed weekend format (iCBT) with a standard group delivery format involving 3 months of weekly sessions (sCBT). A treatment as usual (TAU) condition will be included to compare outcomes. Veterans with one or more anxiety-based disorder(s) (with or without co-occurring depression) will be randomized to one of the three treatment arms. Veterans will be asked to attend a total of four assessments during the study including a baseline evaluation, 1-month, 3-month, and 6-month follow-ups. Qualitative interviews will be conducted with Veterans who completed iCBT and family members.

ELIGIBILITY:
Inclusion Criteria:

* Veterans enrolled to receive VA medical care
* Current diagnosis of at least one anxiety-based disorder
* Moderate-to-poor life enjoyment and satisfaction
* Stable on psychotropic medication 4 weeks prior to participation
* Willing to be randomized to treatment condition

Exclusion Criteria:

* Active symptoms of mania or psychosis at baseline
* Depression with active suicidal ideation/intent
* Moderate-to-severe cognitive impairment
* Active drug/alcohol abuse during initial 3 months of study enrollment
* Undergoing concurrent transdiagnostic CBT for anxiety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Teng, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans at the Michael E. DeBakey VA Medical Center and affiliated community based outpatient clinics were enrolled in this study from 08/1/2018 to 05/31/2021. Veterans were recruited through direct referrals and advertisements.
Pre-assignment Details: Enrolled participants were excluded from the study prior to randomization if they did not meet study inclusion criteria.
Groups:
- iCBT (Intensive Cognitive Behavioral Therapy): Patients in this arm will receive transdiagnostic CBT delivered in an intensive format over one weekend.
  Intensive Cognitive Behavior Therapy (iCBT): Participants randomized to iCBT will receive 16 hours of cognitive behavioral therapy for anxiety over one weekend. The treatment entails psychoeducation, cognitive restructuring and exposure exercises.
- sCBT (Standard Cognitive Behavioral Therapy): Patients in this arm will receive transdiagnostic CBT delivered in a standard weekly format for 12 weeks.
  Standard Cognitive Behavior Therapy (sCBT): Participants randomized to sCBT will receive 16 hours of cognitive behavioral therapy for anxiety weekly over a period of 12 weeks. The treatment entails psychoeducation, cognitive restructuring and exposure exercises.
- TAU (Treatment as Usual): Patients in this arm will not receive transdiagnostic CBT but will receive treatment as usual.
Period: Enrolled and Randomized
Arm/Group | iCBT (Intensive Cognitive Behavioral Therapy) | sCBT (Standard Cognitive Behavioral Therapy) | TAU (Treatment as Usual)
Started (Participants enrolled and randomized to a treatment condition.) | 99 | 99 | 67
Completed (Participants who started treatment.) | 69 | 79 | 67 (These individuals may have received standard care.)
Not Completed | 30 | 20 | 0
Period: Treatment
Arm/Group | iCBT (Intensive Cognitive Behavioral Therapy) | sCBT (Standard Cognitive Behavioral Therapy) | TAU (Treatment as Usual)
Started (Participants who started treatment.) | 69 | 79 | 67
Completed (Participants who completed treatment.) | 66 | 55 | 67
Not Completed | 3 | 24 | 0
Not completed — Urgent Family Matters | 3 | 0 | 0
Not completed — Scheduling Conflicts | 0 | 11 | 0
Not completed — No Longer Interested | 0 | 12 | 0
Not completed — Transportation Issues | 0 | 1 | 0
Period: 1 Month Follow-Up
Arm/Group | iCBT (Intensive Cognitive Behavioral Therapy) | sCBT (Standard Cognitive Behavioral Therapy) | TAU (Treatment as Usual)
Started (Participants who completed treatment.) | 66 | 55 | 67
Completed (Participants who completed 1-Month Follow-Up.) | 57 | 51 | 51
Not Completed | 9 | 4 | 16
Not completed — Lost to Follow-up | 7 | 4 | 15
Not completed — Relocated to Different State | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: 3 Month Follow-Up
Arm/Group | iCBT (Intensive Cognitive Behavioral Therapy) | sCBT (Standard Cognitive Behavioral Therapy) | TAU (Treatment as Usual)
Started | 66 | 55 | 67
Completed | 54 | 44 | 53
Not Completed | 12 | 11 | 14
Not completed — Lost to Follow-up | 11 | 11 | 14
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: 6 Month Follow-Up
Arm/Group | iCBT (Intensive Cognitive Behavioral Therapy) | sCBT (Standard Cognitive Behavioral Therapy) | TAU (Treatment as Usual)
Started | 66 | 55 | 67
Completed | 53 | 46 | 49
Not Completed | 13 | 9 | 18
Not completed — Lost to Follow-up | 12 | 9 | 18
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One participant randomized to the sCBT arm was excluded from analyses due to not meeting study inclusion criteria.
Groups:
- TAU (Treatment a Usual): Patients in this arm will not receive transdiagnostic CBT but will receive treatment as usual.
- Total: Total of all reporting groups
Arm/Group | iCBT (Intensive Cognitive Behavioral Therapy) | sCBT (Standard Cognitive Behavioral Therapy) | TAU (Treatment a Usual) | Total
Number analyzed (Participants) | 99 | 98 | 67 | 264
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.7 (11.2) | 43.9 (12.2) | 43.6 (11.9) | 43.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 34 | 23 | 92
  Male | 64 | 64 | 44 | 172
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 24 | 14 | 63
  Not Hispanic or Latino | 73 | 72 | 50 | 195
  Unknown or Not Reported | 1 | 2 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 0 | 4
  Asian | 2 | 3 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 6 | 1 | 0 | 7
  Black or African American | 46 | 46 | 37 | 129
  White | 35 | 36 | 24 | 95
  More than one race | 5 | 6 | 2 | 13
  Unknown or Not Reported | 3 | 4 | 4 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 99 | 98 | 67 | 264

OUTCOME MEASURES:

1. Primary Outcome: CRIS-EPS: Comparison of Extent of Participation Scores Among iCBT, sCBT, and TAU Groups From Baseline to 1, 3, and 6 Month Follow Ups
Description: The Community Reintegration of Service Members (CRIS) is a commonly used measure of community reintegration in service members and participation in life roles following deployment. The Extent of Participation Subscale (EPS) asks how often an individual experiences/participates in specific activities. Scores on this subscale range from 1 - 7, with higher scores indicating greater degrees of participation in life roles.
Time Frame: Baseline, 1 Month, 3 Month, 6 Month Follow Ups
Population: The number of participants reported here differ from the numbers reported in the Participant Flow because some participants did not complete follow-up assessments at all time points. Also, some participants who completed a follow-up at a later time may not have completed a follow-up at an earlier time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iCBT (Intensive Cognitive Behavioral Therapy) | sCBT (Standard Cognitive Behavioral Therapy) | TAU (Treatment as Usual)
Number analyzed (Participants) | 99 | 98 | 67
score on a scale
  Baseline | 4.21 (0.7) | 4.18 (0.6) | 4.17 (0.8)
  1 Month Follow Up | 4.52 (0.9) | 4.44 (.8) | 4.18 (0.8)
  3 Month Follow Up: number analyzed (Participants) | 53 | 41 | 67
  3 Month Follow Up | 4.57 (.7) | 4.54 (.9) | 4.34 (0.8)
  6 Month Follow Up: number analyzed (Participants) | 53 | 44 | 48
  6 Month Follow Up | 4.70 (0.7) | 4.52 (0.8) | 4.36 (0.8)

2. Primary Outcome: CRIS-PLS: Comparison of Perceived Limitation Scores Among iCBT, sCBT, and TAU Groups From Baseline to 1, 3, and 6 Month Follow Ups
Description: The Community Reintegration in Service Members (CRIS) scale is a commonly used measure of community reintegration in service members and participation in life roles following deployment. The Perceived Limitations Subscale (PLS) asks an individual their perceived limitations in participation. Scores on this subscale range from 1 - 7, with higher scores indicating fewer limitations in participation.
Time Frame: Baseline, 1 Month, 3 Month, 6 Month Follow Ups
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iCBT (Intensive Cognitive Behavioral Therapy) | sCBT (Standard Cognitive Behavioral Therapy) | TAU (Treatment as Usual)
Number analyzed (Participants) | 99 | 98 | 67
score on a scale
  Baseline | 4.40 (0.8) | 4.34 (0.7) | 4.36 (0.9)
  1 Month Follow Up: number analyzed (Participants) | 56 | 50 | 51
  1 Month Follow Up | 4.52 (0.9) | 4.44 (0.8) | 4.18 (0.8)
  3 Month Follow Up: number analyzed (Participants) | 53 | 41 | 51
  3 Month Follow Up | 4.86 (0.9) | 4.52 (0.9) | 4.40 (0.9)
  6 Month Follow Up: number analyzed (Participants) | 53 | 44 | 48
  6 Month Follow Up | 4.70 (0.7) | 4.52 (0.8) | 4.36 (0.8)

3. Primary Outcome: CRIS-SPS: Comparison of Satisfaction With Participation Scores Among iCBT, sCBT, and TAU Groups From Baseline to 1, 3, and 6 Month Follow Ups
Description: The Community Reintegration Service Members (CRIS) scale is a commonly used measure of community reintegration in service members and participation in life roles following deployment. The Satisfaction with Participation Subscale (SPS) asks an individual their degree of satisfaction with participation. Scores on this subscale range from 1 - 7, with higher scores indicating greater levels of satisfaction with their participation.
Time Frame: Baseline, 1 Month, 3 Month, 6 Month Follow Ups
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iCBT (Intensive Cognitive Behavioral Therapy) | sCBT (Standard Cognitive Behavioral Therapy) | TAU (Treatment as Usual)
Number analyzed (Participants) | 99 | 98 | 67
score on a scale
  Baseline | 4.28 (1.0) | 4.26 (1.2) | 4.15 (1.0)
  1 Month Follow Up: number analyzed (Participants) | 56 | 50 | 51
  1 Month Follow Up | 4.80 (1.1) | 4.51 (1.0) | 4.31 (1.0)
  3 Month Follow Up: number analyzed (Participants) | 53 | 41 | 51
  3 Month Follow Up | 4.86 (0.9) | 4.60 (1.0) | 4.40 (0.9)
  6 Month Follow Up: number analyzed (Participants) | 53 | 43 | 47
  6 Month Follow Up | 4.96 (0.8) | 4.63 (1.0) | 4.45 (0.9)

4. Primary Outcome: BAI: Comparison of Beck Anxiety Inventory Scores Among iCBT, sCBT, and TAU Groups From Baseline to 1, 3, and 6 Month Follow Ups
Description: The Beck Anxiety Inventory (BAI) assesses the severity of anxiety symptoms across 21 items, minimizing those that overlap with depression. The BAI assesses cognitive and somatic components of anxiety. The cognitive subscale provides a measure of fearful thoughts and impaired cognitive functioning, whereas the somatic subscale measures the symptoms of physiological arousal. The total score on the BAI ranges from 0 - 63, with higher scores reflecting higher levels of anxiety.
Time Frame: Baseline, 1 Month, 3 Month, 6 Month Follow Ups
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iCBT (Intensive Cognitive Behavioral Therapy) | sCBT (Standard Cognitive Behavioral Therapy) | TAU (Treatment as Usual)
Number analyzed (Participants) | 99 | 98 | 67
score on a scale
  Baseline | 31.8 (11.2) | 31.7 (10.9) | 32.0 (12.1)
  1 Month Follow Up | 24.0 (12.6) | 25.9 (10.3) | 26.3 (12.6)
  3 Month Follow Up: number analyzed (Participants) | 54 | 43 | 53
  3 Month Follow Up | 24.3 (12.2) | 25.6 (11.8) | 26.7 (12.4)
  6 Month Follow Up: number analyzed (Participants) | 53 | 45 | 49
  6 Month Follow Up | 21.6 (11.6) | 24.1 (11.4) | 27.0 (12.1)

5. Secondary Outcome: QLES-SF: Comparison of Quality of Life Enjoyment and Satisfaction Scores Among iCBT, sCBT, and TAU Groups From Baseline to 1, 3, and 6 Month Follow Ups
Description: The Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (QLES-Q-SF) measures subjective functioning and satisfaction across a range of life domains including work, leisure activities, social relationships, and physical health. Satisfaction scores on this measure range from 14 (very poor) to 70 (very good). Higher scores indicate greater overall life satisfaction/functioning.
Time Frame: Baseline, 1 Month, 3 Month, 6 Month Follow Ups
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iCBT (Intensive Cognitive Behavioral Therapy) | sCBT (Standard Cognitive Behavioral Therapy) | TAU (Treatment as Usual)
Number analyzed (Participants) | 99 | 98 | 67
score on a scale
  Baseline | 34.4 (7.0) | 34.8 (5.5) | 33.6 (7.0)
  1 Month Follow Up | 42.9 (9.7) | 40.7 (8.4) | 37.4 (8.3)
  3 Month Follow Up: number analyzed (Participants) | 54 | 54 | 53
  3 Month Follow Up | 42.9 (10.6) | 42.0 (8.9) | 38.3 (9.6)
  6 Month Follow Up: number analyzed (Participants) | 53 | 45 | 49
  6 Month Follow Up | 43.7 (10.1) | 42.5 (8.8) | 38.0 (8.0)

6. Secondary Outcome: BDI-II: Comparison of Beck Depression Inventory Scores Among iCBT, sCBT, and TAU Groups From Baseline to 1, 3, and 6 Month Follow Ups
Description: The Beck Depression Inventory-II (BDI-II) is a well-validated 21-item measure that assesses symptoms of depression. The total score on the BDI-II ranges from 0 - 63, with higher scores reflecting higher levels of depression.
Time Frame: Baseline, 1 Month, 3 Month, 6 Month Follow Ups
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iCBT (Intensive Cognitive Behavioral Therapy) | sCBT (Standard Cognitive Behavioral Therapy) | TAU (Treatment as Usual)
Number analyzed (Participants) | 99 | 98 | 67
score on a scale
  Baseline | 31.0 (10.7) | 31.0 (10.6) | 32.7 (11.1)
  1 Month Follow Up | 23.5 (13.4) | 24.6 (11.8) | 29.8 (12.9)
  3 Month Follow Up: number analyzed (Participants) | 54 | 43 | 53
  3 Month Follow Up | 25.1 (12.7) | 24.8 (13.2) | 28.5 (13.1)
  6 Month Follow Up: number analyzed (Participants) | 53 | 44 | 48
  6 Month Follow Up | 22.5 (12.0) | 24.4 (13.5) | 28.8 (12.8)

ADVERSE EVENTS:
Time Frame: 3 years, 7 months
Description: Adverse events were systematically evaluated throughout the course of the study, from baseline through the last follow-up period. At each time point, medical records for each participant were reviewed and symptoms were monitored through measures administered to each participant. One participant randomized to the sCBT arm was excluded from analyses due to not meeting study inclusion criteria.
Arm/Group | iCBT (Intensive Cognitive Behavioral Therapy) | sCBT (Standard Cognitive Behavioral Therapy) | TAU (Treatment as Usual)
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/98 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/98 | 0/67
Other Adverse Events (participants affected / at risk) | 0/99 | 0/98 | 0/67

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic, all research was placed on hold for several months. All study procedures for this project had to be converted to virtual telehealth delivery. This change in modality (including intervention delivery) may have impacted study outcomes and resulted in underpowered analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT03810456/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT03810456/SAP_001.pdf